CLINICAL TRIAL: NCT07135479
Title: Effects of Youth Mental Health First Aid Training
Brief Title: Effects of Youth Mental Health First Aid (YMHFA) on South Asian American Adults Working With South Asian American Youth
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, College Park (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 1366194
Record Dates: First submitted 2025-08-11; First posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Waitlist Control; Experimental
Keywords: Youth Mental Health First Aid; South Asian American adults; South Asian American youth; South Asian American mental health

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Youth Mental Health First Aid
  Interventions: Other: Youth Mental Health First Aid
- Waitlist Control Group (Active Comparator): Youth Mental Health First Aid
  Interventions: Other: Youth Mental Health First Aid

INTERVENTIONS:
Other: Youth Mental Health First Aid — This Youth Mental Health First Aid training has been adapted for South Asian American adults working with South Asian American youth. This training is a full-day, 5.25 hour blended course (some self-paced work and some live, virtual participation).

SUMMARY:
This study aims to adapt the Youth Mental Health First Aid training to better meet the needs of South Asian American adults who support South Asian American youth. Focus groups will help identify what changes are needed. Based on that input, the training will be updated and then tested to see how well it helps adults improve their knowledge, attitudes, and behaviors toward mental health and supporting the mental health of South Asian American youth.

DETAILED DESCRIPTION:
Youth Mental Health First Aid (YMHFA) USA is a public education program which introduces participants to the unique risk factors and warning signs of mental health problems in adolescents, builds understanding of the importance of early intervention, and teaches individuals how to help an adolescent in crisis or experiencing a mental health challenge. Mental Health First Aid uses role-playing and discussion to demonstrate how to assess a mental health crisis, select interventions and provide initial help, and connect young people to professional, peer, social, and self-help care.

The goal of YMHFA is to ensure everyone in America has at least one First Aider in their close circle of friends, family and peers. Every 1 in 15 people should be certified to identify, understand and respond to signs and symptoms of mental health and substance use challenges.

Though YMHFA has trained more than 4 million First Aiders and there is ample research done on how the training can improve knowledge, attitudes, and behaviors of those working with youth, little to no research has demonstrated the impacts of the training for South Asian American (SAA) adults working with SAA youth.

This project is investigating the cultural adaptation of YMHFA for the SAA community, specifically looking to reflect the values and perspectives embedded within the culture/community, challenges SAA youth are experiencing, and the various cultural factors/considerations that may facilitate/hinder help-seeking when needed. This information will be gathered by conducting focus groups with SAA adults and SAA youth to understand their experiences, how one conceptualizes mental health, what challenges they have experienced or observed, and seek their feedback on some aspects of the training for adaptation consideration. Upon completion of the focus groups, the transcripts will be reviewed and thematized to inform the final adaptations implemented.

Additionally, survey data will be collected from participants before and one month after completing the training to better understand how the adapted training may improve mental health knowledge, help-seeking attitudes and behaviors, and the utilization of the skills taught within the training for SAA adults working with SAA youth.

The findings will provide implications for the role cultural adaptation may play for YMHFA and other mental health/well-being trainings. Moreover, the findings can help to shed light on ways in which we can better approach this community and SAA youth when it comes to mental health conversations, supporting their needs, and encouraging professional and/or informal support. Finally, we hope the adaptations identified can inform additional tools and resources the National Council for Mental Wellbeing may provide to YMHFA instructors who may also train other SAA individuals/communities/organizations.

ELIGIBILITY:
Inclusion Criteria:

* South Asian American adults (18+) working with South Asian American youth (between 8-18 years old)
* Have not taken and completed YMHFA training before

Exclusion Criteria:

* Identify outside of being a South Asian American adult (18+)
* Have taken and completed YMHFA training before
* Mental health professionals/those with a mental health background

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2025-06-24 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Mental Health Literacy Scale (MHLS) | From enrollment to before participating in the Youth Mental Health First Aid (YMHFA) training and one month after participating in the YMHFA training.
  The Mental Health Literacy Scale (MHLS) is a 35-item tool that assesses knowledge across a variety of domains related to mental health, including attitudes toward mental health and help-seeking behaviors. Items 1 to 10 and 13 to 15 are rated on a 4-point Likert scale from 1 (very unlikely) to 4 (very likely). Items 11 to 12 are rated on 4-point Likert scale ranging from 1 (very unhelpful) to 4 (very helpful). Additionally, items 16 to 28 are rated on 5-point Likert scale ranging from 1 (strongly disagree) to 5 (strongly agree), with items 29 to 35 also rated on 5-point Likert scale ranging from 1 (definitely unwilling) to 4 (definitely willing). Overall, higher total scores indicate greater mental health literacy (better outcome).
Confidence in Helping Skills | From enrollment to before participating in the YMHFA training and one month after participating in the YMHFA training.
  The "Confidence in Helping Skills" 5-item measure will assess adults' confidence in applying the ALGEE steps (part of YMHFA training). Participants will indicate their level of agreement with each statement on a 5-point Likert scale ranging from 1 (strongly disagree) to 5 (strongly agree). Overall, higher scores indicate higher confidence in applying the ALGEE steps (better outcome).
Intentions to engage in Mental Health First Aid behaviors | From enrollment to before participating in the YMHFA training and one month after participating in the YMHFA training.
  Participants' intentions to engage in ALGEE will be measured using responses to two vignettes featuring a youth with depression and another with schizophrenia.
  The responses will be coded using a checklist that scores each ALGEE action step using a 3-point scale from 0 (no mention or inadequate response) to 2 (specific details/actions). Overall, higher scores indicate greater intentions to engage in ALGEE (better outcome).
Mental Health Service Use (MHSU) | From enrollment to before participating in the YMHFA training and one month after participating in the YMHFA training.
  The Mental Health Service Use (MHSU) questionnaire will assess participants' utilization of mental health services within the past month, gauging the frequency of accessing these services for themselves and/or a family member. This scale consists of 9 items on a 6-point Likert scale ranging from 0 days accessing services to more than 10 days accessing services. Overall, the higher the score, the more services that have been accessed by participants (better outcome).
Engagement in MHFA behaviors (ALGEE) | From enrollment to before participating in the YMHFA training and one month after participating in the YMHFA training.
  Engagement in actual MHFA behaviors (ALGEE) will be assessed through participants rating the frequency of their engagement in each ALGEE behavior on a 4-point Likert scale from 1 (never) to 4 (many times). Overall, higher the score indicates participants have engaged in ALGEE behaviors more often (better outcome).
Depression Anxiety Stress Scale (DASS-21) | From enrollment to before participating in the YMHFA training and one month after participating in the YMHFA training.
  Depression Anxiety Stress Scale (DASS-21) consists of 21 items across three subscales that measure symptoms of depression, anxiety, and stress. Participants rate the extent to which they experienced these symptoms over the past week on a scale from 0 (did not apply to me at all) to 3 (applied to me very much or most of the time). Overall, higher the score indicates greater symptom severity for participants (worse outcome).
Barriers to Access to Care Evaluation (BACE v3) | From enrollment to before participating in the YMHFA training and one month after participating in the YMHFA training.
  The Barriers to Access to Care Evaluation (BACE v3) will assess barriers to mental health service utilization. The 30-item measure examines three categories of barriers; however, this study will focus on two categories of barriers (22 items): (1) stigma-related barriers and (2) attitudinal barriers. Each item represents a specific barrier that may have prevented, delayed, or discouraged individuals from seeking professional mental health care. Responses are rated on a 4-point Likert scale ranging from 0 (not at all) to 3 (a lot), with six items including an additional "not applicable" option. Overall, higher scores indicate the more barriers participants faced that may have prevented, delayed, or discouraged them from seeking professional mental health care (worse outcome).

SECONDARY OUTCOMES:
Acceptability | This will only be collected one month after participating in the YMHFA training.
  Satisfaction with the YMHFA training will be assessed using a five-item intervention acceptability scale. Participants will rate these items on a 5-point Likert scale from 1 (strongly disagree) to 5 (strongly agree). Overall, higher the score indicates a greater acceptability of the training (better outcome).

CONTACTS AND LOCATIONS:
Overall Officials: Cixin Wang, Ph.D., Study Chair — University of Maryland, College Park
Locations (1):
- UMD College of Education, College Park, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2025-06-20): https://cdn.clinicaltrials.gov/large-docs/79/NCT07135479/ICF_000.pdf